CLINICAL TRIAL: NCT00074399
Title: Nevirapine (NVP) Use to Prevent Maternal-Infant HIV Transmission: A Randomized Clinical Trial of Two Doses of NVP Compared to Six Weeks of NVP for the Prevention of Maternal-Infant HIV Transmission in the Breastfeeding Infant
Brief Title: Nevirapine (NVP) Use to Prevent Mother-to-Child Transmission of HIV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Elham Hassen, MD, Johns Hopkins University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 5R01AI038576-05 (NIH); NIGAT Project
Record Dates: First submitted 2003-12-11; First posted 2003-12-15 (Estimated); Last update posted 2009-08-07 (Estimated); Status verified 2009-08

CONDITIONS: HIV Infections
Keywords: Maternal/Infant Transmisson; Vertical Transmission; Pregnancy; HIV Seronegativity
MeSH Terms: conditions — HIV Infections | interventions — Nevirapine

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- 1 (Experimental): Participants will receive nevirapine for 6 weeks
  Interventions: Drug: Nevirapine
- 2 (Placebo Comparator): Participants will receive nevirapine placebo for 6 weeks
  Interventions: Drug: Nevirapine placebo

INTERVENTIONS:
Drug: Nevirapine — Tablet taken orally daily. Dosage depends on age and body surface area
  Arms: 1
Drug: Nevirapine placebo — Placebo tablet taken orally daily
  Arms: 2

SUMMARY:
HIV can be transmitted from an HIV infected mother to her infant through her breast milk. The purpose of this study is to determine whether giving infants of HIV infected mothers the anti-HIV drug nevirapine (NVP) for six weeks will reduce the risk of HIV transmission.

Study hypothesis: Six weeks of nevirapine prophylaxis provided to the infant will decrease HIV transmission through breastfeeding.

DETAILED DESCRIPTION:
The use of antiretroviral therapy during late pregnancy, intrapartum, and immediately postpartum prevents a high proportion of vertical transmission. Potential means of decreasing HIV transmission through breastfeeding, along with the risks and benefits of early weaning, need to be further evaluated. The potential impact of early weaning interventions on the breastfeeding habits of the HIV uninfected population needs to be considered as well. This study seeks to identify a way to make breastfeeding safe for HIV infected women who choose to breastfeed.

A single dose of NVP given to infants of HIV infected mothers appears to provide some protection against vertical transmission. NVP's long half-life allows simple dosing, making it more feasible and affordable to implement in a developing country. This study will determine whether extending the NVP dosing to six weeks will significantly decrease transmission during the first several months of breastfeeding.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection, documented on two separate specimens
* Estimated gestational age at enrollment of 32 weeks or more as indicated by last menstrual cycle and fundal height
* Permanent residency in Addis Ababa
* Plan to deliver at a hospital affliated with the study (Tikur Anbessa Hospital, Gandhi hospital, or St. Paul's Hospital)
* Hemoglobin >= 7.5 gm/dl within 4 weeks prior to study entry
* Serum glutamic pyruvic transaminase (SGPT) < 5 times upper limit of normal within 4 weeks prior to study entry
* Serum creatinine < 1.5 mg/dl within 4 weeks prior to study entry
* Consent form signed by the mother and, when possible, by the father, prior to the onset of labor

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 775 (Actual)
Dates: Start 2001-02; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Infant HIV infection status | At Months 6 and 12

SECONDARY OUTCOMES:
Infant mortality rate | Throughout study
Infant morbidity rate | Throughout study

CONTACTS AND LOCATIONS:
Locations (1):
- Tikur Anbessa Hospital, Addis Ababa, Ethiopia

REFERENCES:
- [Derived] Six Week Extended-Dose Nevirapine (SWEN) Study Team; Bedri A, Gudetta B, Isehak A, Kumbi S, Lulseged S, Mengistu Y, Bhore AV, Bhosale R, Varadhrajan V, Gupte N, Sastry J, Suryavanshi N, Tripathy S, Mmiro F, Mubiru M, Onyango C, Taylor A, Musoke P, Nakabiito C, Abashawl A, Adamu R, Antelman G, Bollinger RC, Bright P, Chaudhary MA, Coberly J, Guay L, Fowler MG, Gupta A, Hassen E, Jackson JB, Moulton LH, Nayak U, Omer SB, Propper L, Ram M, Rexroad V, Ruff AJ, Shankar A, Zwerski S. Extended-dose nevirapine to 6 weeks of age for infants to prevent HIV transmission via breastfeeding in Ethiopia, India, and Uganda: an analysis of three randomised controlled trials. Lancet. 2008 Jul 26;372(9635):300-13. doi: 10.1016/S0140-6736(08)61114-9. PMID 18657709